CLINICAL TRIAL: NCT06703697
Title: Evaluating the Effectiveness and Implementation of Mobile Health Platform for Medication Management and E-Labeling (eDrugSafe): a Cluster Randomized Trial
Brief Title: Effectiveness and Implementation of Mobile Health Platform for Medication Management and E-Labeling (eDrugSafe)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Jung Mi Oh, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SNUH IRB 2403_002-015; 22183MFDS499 (Other Grant/Funding Number: Ministry of Food and Drug Safety (MFDS), Republic of Korea)
Record Dates: First submitted 2024-11-06; First posted 2024-11-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Mobile Health; Medication Management; Drug Labelling
Keywords: Mobile Health; Medication Management; Drug E-label; electronic labeling; hybrid study; implementation; cluster randomized trial; Electronic Medicinal Product Information (ePI)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: eDrugSafe (Experimental): Participants will use the eDrugSafe mobile web platform to manage their medication history and access electronic medicinal product information (ePI). QR codes are provided with each prescription to connect users directly to ePI content.
  Interventions: Other: eDrugSafe
- Control group: Usual care (No Intervention): Participants will use traditional methods, like paper, for managing and accessing medication information. Use of any digital platforms is not permitted in this group.

INTERVENTIONS:
Other: eDrugSafe — The eDrugSafe mobile web platform enables management of medication history and provides electronic access to medicinal product information (ePI). QR codes are separately provided for prescription records to facilitate direct access to ePI.
  Other Names: eDrugSafe: mobile web platform
  Arms: Intervention group: eDrugSafe

SUMMARY:
The goal of this cluster randomized trial is to learn if eDrugSafe, a mobile web platform for drug electronic labeling (e-labeling) and medication management, can improve medication adherence and self-efficacy in adults who take multiple medications. This study will also assess whether eDrugSafe is feasible and acceptable for use in real clinical settings, especially in local pharmacies.

The main questions it aims to answer are:

* Can eDrugSafe improve medication adherence, self-efficacy, and quality of life for adults taking multiple medications and reduce hospitalizations?
* Is eDrugSafe acceptable and feasible for implementing drug e-labeling and supporting medication management in community settings?

Researchers will compare eDrugSafe to usual care (traditional paper methods) to see if eDrugSafe is effective in supporting adults who take multiple medications, and if it can be feasibly implemented in local pharmacies.

Participants will:

* Visit a local pharmacy randomly assigned to use eDrugSafe or traditional care methods and decide if they wish to join the study.
* Use either eDrugSafe to access medication information and manage their medication history, or receive usual care with paper-based methods, for 6 months.
* Complete surveys at the start of the study, at 3 months, and at 6 months to measure effectiveness and implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 79 years.
2. Individuals who can speak and understand Korean.
3. Possession of a personal electronic device capable of accessing mobile applications and web services over wireless internet (bring participants' own device, BYOD).
4. Patients taking three or more medications with at least one medication prescribed for 28 days or longer.
5. Individuals who have provided direct consent to participate in the study.

Exclusion Criteria:

1. Individuals using any mobile web platform other than eDrugSafe for medication safety information purposes after enrollment.
2. Individuals who do not consent to participate in the study or who withdraw their consent.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: medication adherence | baseline, 3 month, 6 month
  * Assessment: The Korean version of the Morisky Medication Adherence Scale-8 (MMAS-8)
  * Units of Measure: Total MMAS-8 score (range: 0-8)
  * Description: The MMAS-8 scale consists of 8 items. Each of the first 7 items has 2 possible responses (yes/no), while the 8th item is answered with a 5-point Likert scale. The possible total medication adherence score ranges between 0 and 8, and the higher the score, the better the adherence level. A total score < 6 is considered low adherence, while a total score of ≥ 6 but < 8 indicates moderate adherence, and a score of 8 indicates high adherence.
Effectiveness: self-efficacy in medication management | baseline, 3 month, 6 month
  * Assessment: The Korean version of the Self-Efficacy for Appropriate Medication Use Scale (SEAMS)
  * Units of Measure: Total SEAMS score (range: 16-48)
  * Description: The SEAMS is a 16-item scale that assesses confidence in managing medications. Higher scores indicate greater self-efficacy and confidence in medication management.

SECONDARY OUTCOMES:
Effectiveness: Health-related quality of life | 6 month
  * Units of Measure: EQ-5D-5L Index (-1 to 1)
  * Description: Health-related quality of life at the 6-month follow-up will be assessed using the Korean EQ-5D-5L scale, administered electronically. The EQ-5D-5L measures five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on five levels (no problems to extreme problems). Responses are converted to an index value (1: full health to 0: death; below 0: worse than death) using a validated Korean scoring algorithm.
Effectiveness: Health-related quality of life | 6 month
  * Units of Measure: EQ-5D-5L VAS Score (0 to 100)
  * Description: Health-related quality of life at the 6-month follow-up will be assessed using the Korean EQ-5D-5L scale, administered electronically. A Visual Analogue Scale (VAS) will also measure self-rated health on a scale from 0 (worst) to 100 (best), administered concurrently with the EQ-5D-5L.
Effectiveness: Emergency room visits | 6 month
  * Units of Measure: Number of emergency room visits (count)
  * Description: Higher counts reflect poor health outcomes.
Effectiveness: Hospitalizations | 6 month
  * Units of Measure: Number of hospitalizations (count)
  * Description: Higher counts reflect poor health outcomes.

OTHER OUTCOMES:
Implementation: Feasibility of mobile web platform | 6-month follow-up (intervention group only)
  * Assessment: Semi-structured survey guided by the RE-AIM and CFIR frameworks
  * Units of Measure: Descriptive statistics of response frequencies (quantitative data) and qualitative analysis
  * Description: The survey assesses user perspectives across three areas: study background, experience with e-labels and the platform, and potential for adoption. Quantitative data will include descriptive statistics of response frequencies, while qualitative data will be analyzed using word coding to identify themes such as acceptability, adoption, feasibility, and barriers.
Implementation: Usability of mobile web platform | 6-month follow-up (intervention group only)
  * Assessment: Korean System Usability Scale (SUS)
  * Units of Measure: SUS total score (range: 0-100)
  * Description: The SUS is a 10-item tool used to assess the usability of the mobile web platform. Scores range from 0 to 100 and are calculated by adjusting responses and multiplying the total by 2.5. A score above 68 is considered above average for usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
The decision not to share individual participant data is based on the potential inclusion of certain personal information in the research data. Furthermore, informed consent was not obtained from participants for the disclosure of their information to third parties or public databases.